CLINICAL TRIAL: NCT02393053
Title: Innovation Technique With Non-pedicled Buccal Fat Pad Graft in the Treatment of Gingival Recessions: a Randomized Controlled Clinical Trial
Brief Title: Non-Pedicled Buccal Fat Pad Graft in the Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Positivo (Other)
Responsible Party: Principal Investigator, Tatiana Miranda Deliberador, Full Professor, Universidade Positivo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PositivoU
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Case-Control Studies; Adipose Tissue
MeSH Terms: conditions — Gingival Recession | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- subepithelial connective tissue graft (Sham Comparator): Surgery: Treatment with subepithelial connective tissue graft for gingival recession
  Interventions: Procedure: Treatment with subepithelial connective tissue graft (SCTG)
- non-pedicled buccal fat pad graft (Experimental): Surgery: Treatment with non-pedicled buccal fat pad graft for gingival recession
  Interventions: Procedure: Treatment with non-pedicled buccal fat pad graft (BFPG)

INTERVENTIONS:
Procedure: Treatment with subepithelial connective tissue graft (SCTG) — Miller Class I or II gingival recessions were treated with subepithelial connective tissue graft (SCTG)
  Arms: subepithelial connective tissue graft
Procedure: Treatment with non-pedicled buccal fat pad graft (BFPG) — Miller Class I or II gingival recessions were treated with non-pedicled buccal fat pad graft (BFPG)
  Arms: non-pedicled buccal fat pad graft

SUMMARY:
Background: This randomized controlled clinical study of split-mouth aimed to compare non-pedicled buccal fat pad graft (BFPG) with subepithelial connective tissue graft (SCTG) in the treatment of Miller Class I or II gingival recessions.

Methods: Twelve patients with Miller Class I or II (≥ 2 mm) bilateral recessions in maxillary premolars or canines were selected. The recessions were randomly assigned to receive SCTG (Control Group) or BFPG (Test Group). The clinical parameters of Gingival Index (GI), Plaque Index (PI), Probing Depth (PD), Gingival Recession (GR), Clinical Attachment Level (CAL), Width of Keratinized Tissue (WKT), Thickness of Keratinized Tissue (TKT) and Gingival Margin to the Acrylic Guide (GM-AG) were evaluated at baseline, and in the postoperative periods of 1, 3, and 6 months. The percentage of root coverage was also evaluated. Data were submitted to repeated measures ANOVA, Bonferroni method and t-test (p<0.05).

DETAILED DESCRIPTION:
MATERIALS AND METHODS

Study population This paper aims to report a randomized controlled clinical study of split-mouth. 12 patients were selected, 8 women and 4 men, aged between 21 and 65 (mean age 41 ± 11.9 years). They were informed about the risks and benefits of this clinical investigation as well as associated procedures, and signed a free and informed consent form. This study was approved by the Ethics and Research Committee of Positivo University (083/2010).

The inclusion criteria for the selection of patients were: 1) patients with Miller Class I or II gingival recessions located bilaterally in the vestibular surface of upper premolars or canines ≥ to 2 mm; 2) patients who had recessions with some differences between the right and the left sides ≤ to 3 mm; 3) non-smokers; 4) non-pregnant patients; 5) systemically healthy patients; 6) periodontally healthy patients with no contraindications for periodontal surgery; 7) patients who did not take any kind of medicine that could interfere with the health of gingival and periodontal tissue; 8) teeth with probing depth (PD) <3 mm and without bleeding on probing (BOP); 9) teeth with no caries or restorations in the cervical region; and 10) region that had not been undergone any periodontal surgery before.

Initial therapy The patients underwent a basic periodontal treatment including scaling, root planing, tooth polishing and oral hygiene instructions as required. Additionally, all patients were included in a pre-treatment program in order to eliminate possible etiological factors related to gingival recession. Patients were instructed to perform a non-traumatic brushing technique by using a toothbrush with soft bristles. The surgical procedure was performed only in patients who had adequate plaque control.

Clinical Parameters After 30 days of initial therapy, the clinical parameters were recorded by a single calibrated operator with professional experience in periodontics, at the beginning (baseline), and in the postoperative periods of 1, 3, and 6 months respectively. The periodontal probe used was North Carolina (UNC-15, Hu-Friedy, Chicago, IL, USA).

At baseline, an acrylic resin guide was made directly in the mouth of each patient and in each experimental tooth. A reference point (slot) was created in the most central vestibular portion of the guide in order to obtain a fixed reproduction of the periodontal probe position so that the measures of the clinical parameters could be standardized.

The clinical parameters evaluated were: Gingival Index (GI)16; Plaque Index (PI)17; Probing Depth (PD) - measure from the gingival margin (GM) up to the bottom of the gingival sulcus; Gingival Recession (GR) - measure from the Cemento-Enamel Junction (CEJ) up to the GM; Clinical Attachment Level (CAL) - measure from the CEJ up to the bottom of the gingival sulcus; Width of Keratinized Tissue (WKT) - measure from the Mucogingival Junction (MGJ) up to the GM; Thickness of Keratinized Tissue (TKT) - measure performed with the aid of a North Carolina periodontal probe (UNC-15, Hu-Friedy, Chicago, IL, USA) perpendicularly placed along the tooth axis in the most central portion of the keratinized tissue, between the GM and the MGJ. The probe was slightly pressured, under local anesthetic, towards the adjacent hard tissue. Then, the measure in millimeters was recorded and the last mean calculated referred to the Gingival Margin to the Acrylic Guide (GM-AG) - measure performed from the GM up to the most coronal point of the acrylic resin guide.

Surgical Procedure All surgical procedures were performed by the same operator, experienced and specialist in Periodontics. The bilateral gingival recessions were randomly assigned by lot (by a flip of coins) for both the side that received the SCTG (Control Group - C) and the side that received the BFPG (Test Group - T). The same operator performed both surgeries on the same day.

Before the surgical procedure, extra intra-oral antisepsis was performed with 0.12% chlorhexidine digluconate. The clinical parameters GI and PI were evaluated. Then, measures of the clinical parameters PD, GR, CAL, WKT and GM-AG were performed with the aid of an acrylic guide.

Preparation of the recipient site After local infiltration anesthetic (mepivacaine HCL 2% + epinephrine 1:100,000) at the bottom of the vestibule in the region of the upper canine or upper premolar teeth, the measure TKT was performed. Then, an intrasulcular incision was made with a scalpel blade no 15c from the distal side of the upper canine tooth or the premolar tooth towards their mesial side, with great care so that the interdental papillae could be preserved. After that, two divergent vertical releasing incisions were made towards the bottom of the vestibule. A partial-thickness flap was raised releasing all muscle fibers so that the flap could be loose to be slid coronally. The roots were gently debrided and flattened with Gracey curettes 5-6 (Hu-Friedy - USA), and the area was rinsed with sterile saline solution for the total removal of dentine debris. Then, with the aid of an acrylic guide, the measure of the most coronal portion of the recipient site to the acrylic guide (CPRS-AG) was performed. The flap had to be raised so that the measure of the most coronal portion of bone tissue over the root to the acrylic guide could be made.

The standard surgical procedure was to start on the patient's right side regardless of the group that would undergo surgery, Group C or Group T. The preparation of the recipient site was conducted the same way for both groups.

Preparation of the donor site In order to obtain connective tissue graft, the patient was given infiltration anesthetic into the hard palate, on the same side of the recipient site randomly chosen by lot to receive the SCTG. The removal of the connective tissue was performed, followed by an L-shaped incision.

Once the graft was harvested, it was immediately positioned onto the recipient site at the level of the CEJ, and fixed through simple sutures in the mesial and distal sides, with a V-shaped compressive suture (Fig. 1A), from the periosteum to the palatine region of the tooth with absorbable suture thread. After the graft was sutured with the aid of an acrylic guide, the following measures were performed: 1) the measure of the most coronal portion of the graft to the acrylic guide (CPG-AG), and 2) the apico-coronal height of the graft (ACHG). The height of the graft ranged from 6.5 to 8.9 mm for all 12 patients.

The flap was positioned coronally in order to cover the connective tissue graft as a whole. Suspensory and simple sutures were made in the releasing incisions with silk thread (Fig. 1B). After the sutures were finished, the measure of the most coronal position of the flap to the acrylic guide (CPF-AG) was performed.

In order to harvest BFPG (Bichat's Ball), a terminal infiltration anesthetic was injected into the region of the upper first and second molars, on the same side of the recipient site that would receive BFPG. A horizontal incision measuring 1.5 cm was made with a blade no.15 at the bottom of the vestibule, in the region of the teeth 16 and 17 or 26 and 27, depending on which side the surgery would be performed in accordance with the random choice established by lot for the Test Group. A curved hemostat was used to divulse the muscles in the spot and to expose the adipose tissue. The Bichat's Ball was exposed as soon as the muscles were divulsed in the spot (Fig. 2A). Then, a small portion of adipose tissue (1.5 cm x 1.5 cm) was removed with the aid of Goldman Fox scissors. After this procedure, the patient's cheek was compressed in order for the wound edges to close, joining the tissue. The donor site was immediately sutured with silk thread 4.0 (Ethicon, Johnson & Johnson A.G., Brazil) through simple stitches.

The BFPG was placed onto the recipient site at the level of the CEJ and fixed through "X"-shaped sutures over the graft (Fig. 2B) with absorbable suture thread (Vicryl 5-0). The same trans-surgical measures that had been performed in the Control Group were also performed in the Test Group. The height of the graft ranged from 7.70 to 10.3 mm for all 12 patients.

The flap was positioned coronally in order to cover the BFPG as a whole. Suspensory and simple sutures were made in the releasing incisions (Fig. 2C). After the sutures were finished, the measure of the most coronal position of the flap to the acrylic guide (CPF-AG) was performed.

Postoperative Protocol The patients were given postoperative instructions, such as: ice compress on the surgical site during the first 04 hours; liquid and/or soft diet for 3 days; the teeth in the surgical region should not be brushed; and the mouth should be rinsed with a mouthwash containing 0.12% chlorhexidine digluconate during 1 minute, every 12 hours for 14 days.

The postoperative medications prescribed were: Amoxicillin 500 mg every 8 hours for 7 days or Clindamycin 300 mg every 8 hours for 7 days to patients allergic to penicillin, and Ibuprofen + arginine 600 mg every 12 hours for 5 days. The sutures were removed 14 days after surgery. After this period, the patients were recommended to gently brush their teeth with a soft-bristle toothbrush.

All patients were included in a monthly program of professional tooth cleaning and oral hygiene instructions, starting on the 30th day until the 180th day after the surgical procedures.

Statistical analysis Repeated Measures ANOVA associated with the Bonferroni method were used to detect inter- and intra-group differences for the clinical parameters PD, GR, CAL, WKT, TKT, and GM-AG. The t-test was used to detect inter-group differences versus time, for the clinical parameters PD, GR, CAL, WKT, TKT, and GM-AG. For the parameters CPRS-AG, CPG-AG, ACHG, and CPF-AG only the t-test was used. The level of significance was 5% for all statistical comparisons. All analyses were made with the aid of the software SPSS Statistics 18.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Miller Class I or II gingival recessions located bilaterally in the vestibular surface of upper premolars or canines ≥ to 2 mm
2. Patients who had recessions with some differences between the right and the left sides ≤ to 3 mm
3. Non-smokers
4. Non-pregnant patients
5. Systemically healthy patients
6. Periodontally healthy patients with no contraindications for periodontal surgery
7. Patients who did not take any kind of medicine that could interfere with the health of gingival and periodontal tissue
8. Teeth with probing depth (PD) <3 mm and without bleeding on probing (BOP)
9. Teeth with no caries or restorations in the cervical region
10. Region that had not been undergone any periodontal surgery before

Exclusion Criteria:

1. Patients who did not meet the inclusion criteria

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) | Baseline, 1, 3, and 6 months respectively
  measure from the gingival margin (GM) up to the bottom of the gingival sulcus
Change in Gingival Recession (GR) | Baseline, 1, 3, and 6 months respectively
  measure from the Cemento-Enamel Junction (CEJ) up to the GM
Change in Clinical Attachment Level (CAL) | Baseline, 1, 3, and 6 months respectively
  measure from the CEJ up to the bottom of the gingival sulcus
Change in Width of Keratinized Tissue (WKT) | Baseline, 1, 3, and 6 months respectively
  measure from the Mucogingival Junction (MGJ) up to the GM
Change in Thickness of Keratinized Tissue (TKT) | Baseline, 1, 3, and 6 months respectively
  measure performed with the aid of a North Carolina periodontal probe (UNC-15, Hu-Friedy, Chicago, IL, USA) perpendicularly placed along the tooth axis in the most central portion of the keratinized tissue, between the GM and the MGJ

CONTACTS AND LOCATIONS:
Overall Officials: Flares Baratto Filho, PhD, Study Chair — Universidade Positivo

REFERENCES:
- [Background] Kassab MM, Badawi H, Dentino AR. Treatment of gingival recession. Dent Clin North Am. 2010 Jan;54(1):129-40. doi: 10.1016/j.cden.2009.08.009. PMID 20103476
- [Background] Zucchelli G, Testori T, De Sanctis M. Clinical and anatomical factors limiting treatment outcomes of gingival recession: a new method to predetermine the line of root coverage. J Periodontol. 2006 Apr;77(4):714-21. doi: 10.1902/jop.2006.050038. PMID 16584355
- [Background] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Background] de Sanctis M, Baldini N, Goracci C, Zucchelli G. Coronally advanced flap associated with a connective tissue graft for the treatment of multiple recession defects in mandibular posterior teeth. Int J Periodontics Restorative Dent. 2011 Nov-Dec;31(6):623-30. PMID 22140664
- [Background] Bittencourt S, Ribeiro Edel P, Sallum EA, Sallum AW, Nociti FH, Casati MZ. Semilunar coronally positioned flap or subepithelial connective tissue graft for the treatment of gingival recession: a 30-month follow-up study. J Periodontol. 2009 Jul;80(7):1076-82. doi: 10.1902/jop.2009.080498. PMID 19563287
- [Background] El Haddad SA, Abd El Razzak MY, El Shall M. Use of pedicled buccal fat pad in root coverage of severe gingival recession defect. J Periodontol. 2008 Jul;79(7):1271-9. doi: 10.1902/jop.2008.070176. PMID 18597611